CLINICAL TRIAL: NCT02813889
Title: SmarToyGym: Smart Detection of Atypical Toy-oriented Actions in At-risk Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 822487; 1R21HD084327-01 (NIH)
Record Dates: First submitted 2016-06-16; First posted 2016-06-27 (Estimated); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy; Developmental Delay; Stroke; Fine Motor Delay; Infant Development; Other Development Delays
Keywords: infant; baby; developmental delay; robotics; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy; Learning Disabilities; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infants (Experimental): Two populations will be involved in testing in the SmarToyGym: 1. Infants exhibiting typical development between 3 months and 11 months of age 2 . Infants exhibiting atypical development (at-risk for neuromotor delay) between 3 months and 11 months of age.
  Interventions: Device: SmarToyGym

INTERVENTIONS:
Device: SmarToyGym — We aim to develop a SmarToyGym where sensitized, wireless toys are strategically hung and placed within reach of infants to elicit toy-oriented body and arm/hand movements. Each toy will be equipped with sensors capable of measuring the infant's grasping actions such as squeezing, pinching, tilting, etc.
  A low-cost 3D motion capture system will be used to collect video data and the infants' reaching and body kinematics in response to the toys. A pressure mat will be used to measure postural changes to detect weight shifts, rolling, crawling and other movements away from the initial posture.

SUMMARY:
The study aims to develop a SmarToyGym where sensitized, wireless toys are strategically hung and placed within reach of infants to elicit toy-oriented body and arm/hand movements. Each toy will be equipped with sensors capable of measuring the infant's grasping actions such as squeezing, pinching, tilting, etc.

A low-cost 3D motion capture system will be used to collect video data and the infants' reaching and body kinematics in response to the toys. A pressure mat will be used to measure postural changes to detect weight shifts, rolling, crawling and other movements away from the initial posture. By capitalizing on these wireless and low-cost technologies, it will permit the regular and non-invasive monitoring of infants, which can lead to detailed, non-obtrusive, quantitative evaluation of motor development. In this vein, the investigators also aim to conduct proof-of-concept testing of the SmarToyGym with atypical and typical developing infants. The investigators will include infants' ages 3 to 11 months who are categorized as high-risk or low-risk using the Bayley Infant Neurodevelopmental Screener.

DETAILED DESCRIPTION:
The proposed research is specifically designed to investigate the ability of a novel tool to identify atypically developing infants from their typically developing peers. Twenty-four infants will be recruited to participate, including 12 who are developing typically and 12 who are identified as at-risk for neuromotor delay. Infants with typical development will be at least 3 months and less than 11 months of age, score in the low-risk category on the Bayley Infant Neurodevelopmental Screener (BINS), score a greater than 85 on all sub-scales of the Bayley Scale of Infant Development (BSID-II), have no history of significant cardiac, orthopedic, or neurological condition, and gestational age at least 37 weeks. Infants at risk for neuromotor delay will be at least 3 months and less than 11 months of age (corrected for preterm birth if applicable), score in the moderate or high risk categories on the BINS, and score an 85 or less on the motor sub-scales of the Bayley Scale of Infant Development (BSID-II). In an effort to decrease variability of the data, infants in each group will be further stratified into an older group (8-10+ months) and a younger group (3-5 months).

ELIGIBILITY:
Inclusion Criteria:

* Infants exhibiting typical development between 3 months and 11 months of age who score in the low-risk category on the Bayley Infant Neurodevelopment Screener (BINS), score greater than 85 on all sub-scales of the Bayley Scale of Infant Development (BSID-II), have no history of significant cardiac, orthopedic or neurological condition and have a gestational age at least 37 weeks.
* Infants exhibiting atypical development (at-risk for neuromotor delay) between 3 months and 11 months of age, score in the moderate or high risk categories on the BINS, and score an 85 or less on the motor sub-scales of the BSID-II.
* Exclusion Criteria:
* Infants outside age range of 3-11 months

Ages: 3 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle J Johnson, PhD, Principal Investigator — Penn Medicine Rittenhouse; Laura Prosser, PT, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Michelle J Johnson, PhD, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lysenko S, Seethapathi N, Prosser L, Kording K, Johnson MJ. Towards Automated Emotion Classification of Atypically and Typically Developing Infants. Proc IEEE RAS EMBS Int Conf Biomed Robot Biomechatron. 2020 Nov-Dec;2020:503-508. doi: 10.1109/BioRob49111.2020.9224271. Epub 2020 Oct 15. PMID 33959406
- [Background] Goyal V, Torres W, Rai R, Shofer F, Bogen D, Bryant P, Prosser L, Johnson MJ. Quantifying infant physical interactions using sensorized toys in a natural play environment. IEEE Int Conf Rehabil Robot. 2017 Jul;2017:882-887. doi: 10.1109/ICORR.2017.8009360. PMID 28813932
- [Background] Shivakumar SS, Loeb H, Bogen DK, Shofer F, Bryant P, Prosser L, Johnson MJ. Stereo 3D tracking of infants in natural play conditions. IEEE Int Conf Rehabil Robot. 2017 Jul;2017:841-846. doi: 10.1109/ICORR.2017.8009353. PMID 28813925
- [Result] Prosser LA, Aguirre MO, Zhao S, Bogen DK, Pierce SR, Nilan KA, Zhang H, Shofer FS, Johnson MJ. Infants at risk for physical disability may be identified by measures of postural control in supine. Pediatr Res. 2022 Apr;91(5):1215-1221. doi: 10.1038/s41390-021-01617-0. Epub 2021 Jun 26. PMID 34175891
- [Result] Chambers C, Seethapathi N, Saluja R, Loeb H, Pierce SR, Bogen DK, Prosser L, Johnson MJ, Kording KP. Computer Vision to Automatically Assess Infant Neuromotor Risk. IEEE Trans Neural Syst Rehabil Eng. 2020 Nov;28(11):2431-2442. doi: 10.1109/TNSRE.2020.3029121. Epub 2020 Nov 6. PMID 33021933
- [Result] Kather C, Shofer FS, Park JI, Bogen D, Pierce SR, Kording K, Nilan KA, Zhang H, Prosser LA, Johnson MJ. Quantifying interaction with robotic toys in pre-term and full-term infants. Front Pediatr. 2023 Oct 19;11:1153841. doi: 10.3389/fped.2023.1153841. eCollection 2023. PMID 37928351

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The same group of infants were analyzed throughout the study and for all outcome measures. The number differs for each outcome measure because data for some infants were excluded, the number varying for each study due to the specific outcome measure. These exclusions are specifically explained for each outcome measure in the outcome measures section. Infants #35 and #36 were consented, but no data was collected for them regarding any outcome measure.
Groups:
- Full-Term Infants; Pre-Term Infants: Two populations will be involved in testing in the SmarToyGym: 1. Full-term infants (born at a gestational age of > 37 weeks) between 3 months and 11 months of age. 2. Pre-term infants (born at a gestational age < 36 weeks) between 3 months and 11 months of age.
  Infants were also categorized by typical and atypical (at-risk for neuromotor delay or physical disability) development.
  SmarToyGym: We aim to develop a SmarToyGym where sensitized, wireless toys are strategically hung and placed within reach of infants to elicit toy-oriented body and arm/hand movements. Each toy will be equipped with sensors capable of measuring the infant's grasping actions such as squeezing, pinching, tilting, etc.
  A low-cost 3D motion capture system will be used to collect video data and the infants' reaching and body kinematics in response to the toys. A pressure mat will be used to measure postural changes to detect weight shifts, rolling, crawling and other movements away from the initial posture.
Period: Overall Study
Arm/Group | Full-Term Infants | Pre-Term Infants
Started | 26 | 10
Completed | 19 | 10
Not Completed | 7 | 0
Not completed — Excluded 7 due to protocol adjustments. Specific exclusions listed under each outcome measure. | 7 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Data were collected from infants irrespective of full term/pre-term status and therefore cannot be separated.
Groups:
- Full-Term and Pre-Term Infants: Two populations will be involved in testing in the SmarToyGym: 1. Full-term infants (born at a gestational age of > 37 weeks) between 3 months and 11 months of age. 2. Pre-term infants (born at a gestational age < 36 weeks) between 3 months and 11 months of age.
  Infants were also categorized by typical and atypical (at-risk for neuromotor delay or physical disability) development, and by low, moderate, and high risk.
  SmarToyGym: We aim to develop a SmarToyGym where sensitized, wireless toys are strategically hung and placed within reach of infants to elicit toy-oriented body and arm/hand movements. Each toy will be equipped with sensors capable of measuring the infant's grasping actions such as squeezing, pinching, tilting, etc.
  A low-cost 3D motion capture system will be used to collect video data and the infants' reaching and body kinematics in response to the toys. A pressure mat will be used to measure postural changes to detect weight shifts, rolling, crawling and other movements away from the initial posture.
Arm/Group | Full-Term and Pre-Term Infants
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: month] | 6 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 21
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Center of Pressure, Path Length Per Second - No Toy (Birth Status)
Description: Body movement (center of pressure) on a mat, in terms of average path length per second. Early postural control (measured by center of pressure) was investigated to distinguish infants with future impairment in motor control from their typically developing peers. Lower path length is representative of greater postural control. The data analyzed was the condition where infant supine movement on the mat for up to two minutes without a toy. Path length was measured in distance with time normalized to 1 minute.
Time Frame: 1 session, about 1 hour in length
Population: 21 excluded from enrolled 36: 7 infants were excluded from Center of Pressure analysis due to procedural adjustments.
  11 infants were excluded from Center of Pressure analysis due to unusable data (infants either rolled or crawled on the mat, or they were fussy and were not able to be calmed while laying supine without being touched).
  3 infants were excluded from Center of Pressure analysis due to technical issues (with the mat on the day of testing).
Measure: Mean (Standard Deviation); unit: centimeters per second (cm/sec)
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 8 | 7
centimeters per second (cm/sec) | 0.0282 (0.0116) | 0.0428 (0.0144)
Statistical Analysis 1: Comparison: Full-Term Infants vs Pre-Term Infants; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.0054, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = -0.0146, 95% CI 2-sided [-0.0261 to -0.0031] — Difference = Path Length (Full-Term) - Path Length (Pre-Term)

2. Primary Outcome: Center of Pressure, Path Length Per Second - Elephant Toy (Birth Status)
Description: Body movement (center of pressure) on a mat, in terms of average path length per second. Early postural control (measured by center of pressure) was investigated to distinguish infants with future impairment in motor control from their typically developing peers. Lower path length is representative of greater postural control. The data analyzed was the condition where infant supine movement on the mat for up to two minutes with elephant toy. Path length was measured in distance with time normalized to 1 minute.
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per second (cm/sec)
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 8 | 7
centimeters per second (cm/sec) | 0.0311 (0.0171) | 0.0508 (0.0206)
Statistical Analysis 1: Comparison: Full-Term Infants vs Pre-Term Infants; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.0005, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = -0.0200, 95% CI 2-sided [-0.0331 to -0.0070] — Difference = Path Length (Full-Term) - Path Length (Pre-Term)

3. Primary Outcome: Center of Pressure, Path Length Per Second - Orangutan Toy (Birth Status)
Description: Body movement (center of pressure) on a mat, in terms of average path length per second. Early postural control (measured by center of pressure) was investigated to distinguish infants with future impairment in motor control from their typically developing peers. Lower path length is representative of greater postural control. The data analyzed was the condition where infant supine movement on the mat for up to two minutes with orangutan toy. Path length was measured in distance with time normalized to 1 minute.
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per second (cm/sec)
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 8 | 7
centimeters per second (cm/sec) | 0.0251 (0.105) | 0.0417 (0.0115)
Statistical Analysis 1: Comparison: Full-Term Infants vs Pre-Term Infants; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.0088, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = -0.0146, 95% CI 2-sided [-0.0267 to -0.0026] — Difference = Path Length (Full-Term) - Path Length (Pre-Term)

4. Primary Outcome: Center of Pressure, Path Length Per Second - Lion Toy (Birth Status)
Description: Body movement (center of pressure) on a mat, in terms of average path length per second. Early postural control (measured by center of pressure) was investigated to distinguish infants with future impairment in motor control from their typically developing peers. Lower path length is representative of greater postural control. The data analyzed was the condition where infant supine movement on the mat for up to two minutes with lion toy. Path length was measured in distance with time normalized to 1 minute.
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per second (cm/sec)
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 8 | 7
centimeters per second (cm/sec) | 0.0342 (0.0123) | 0.0421 (0.0126)
Statistical Analysis 1: Comparison: Full-Term Infants vs Pre-Term Infants; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.7624, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = -0.0059, 95% CI 2-sided [-0.0180 to 0.0062] — Difference = Path Length (Full-Term) - Path Length (Pre-Term)

5. Primary Outcome: Center of Pressure, Path Length Per Second - No Toy (Motor Control Outcome)
Description: Body movement (center of pressure) on a mat, in terms of path length per minute. Early postural control (measured by center of pressure) was investigated to distinguish infants with future impairment in motor control from their typically developing peers. Lower path length is representative of greater postural control. The data analyzed was the condition where infant supine movement on the mat for up to two minutes without a toy. Path length was measured in distance with time normalized to 1 minute.
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per second (cm/sec)
Groups:
- Infants - Typical Development; Infants - Atypical Development: Two populations will be involved in testing in the SmarToyGym: 1. Full-term infants (born at a gestational age of > 37 weeks) between 3 months and 11 months of age. 2. Pre-term infants (born at a gestational age < 36 weeks) between 3 months and 11 months of age.
  Infants were also categorized by typical and atypical (at-risk for neuromotor delay or physical disability) development.
  SmarToyGym: We aim to develop a SmarToyGym where sensitized, wireless toys are strategically hung and placed within reach of infants to elicit toy-oriented body and arm/hand movements. Each toy will be equipped with sensors capable of measuring the infant's grasping actions such as squeezing, pinching, tilting, etc.
  A low-cost 3D motion capture system will be used to collect video data and the infants' reaching and body kinematics in response to the toys. A pressure mat will be used to measure postural changes to detect weight shifts, rolling, crawling and other movements away from the initial posture.
Arm/Group | Infants - Typical Development | Infants - Atypical Development
Number analyzed (Participants) | 11 | 4
centimeters per second (cm/sec) | 0.0287 (0.0110) | 0.0416 (0.0035)
Statistical Analysis 1: Comparison: Infants - Typical Development vs Infants - Atypical Development; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.0326, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = 0.0129, 95% CI 2-sided [0.0007 to 0.0251] — Difference = Path Length per second (Typical) - Path Length per second (Atypical)

6. Primary Outcome: Center of Pressure, Path Length Per Second - Elephant Toy (Motor Control Outcome)
Description: Body movement (center of pressure) on a mat, in terms of path length per minute. Early postural control (measured by center of pressure) was investigated to distinguish infants with future impairment in motor control from their typically developing peers. Lower path length is representative of greater postural control. The data analyzed was the condition where infant supine movement on the mat for up to two minutes with elephant toy. Path length was measured in distance with time normalized to 1 minute.
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per second (cm/sec)
Arm/Group | Infants - Typical Development | Infants - Atypical Development
Number analyzed (Participants) | 11 | 4
centimeters per second (cm/sec) | 0.0312 (0.0153) | 0.0617 (0.0181)
Statistical Analysis 1: Comparison: Infants - Typical Development vs Infants - Atypical Development; Test type: Superiority — Two-Factor ANOVA in repeated measures; p < 0.0001, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = 0.0309, 95% CI 2-sided [0.0138 to 0.0480] — Difference = Path Length per second (Typical) - Path Length per second (Atypical)

7. Primary Outcome: Center of Pressure, Path Length Per Second - Orangutan Toy (Motor Control Outcome)
Description: Body movement (center of pressure) on a mat, in terms of path length per minute. Early postural control (measured by center of pressure) was investigated to distinguish infants with future impairment in motor control from their typically developing peers. Lower path length is representative of greater postural control. The data analyzed was the condition where infant supine movement on the mat for up to two minutes with orangutan toy. Path length was measured in distance with time normalized to 1 minute.
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per second (cm/sec)
Arm/Group | Infants - Typical Development | Infants - Atypical Development
Number analyzed (Participants) | 11 | 4
centimeters per second (cm/sec) | 0.0260 (0.0100) | 0.0445 (0.0070)
Statistical Analysis 1: Comparison: Infants - Typical Development vs Infants - Atypical Development; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.0025, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = 0.0170, 95% CI 2-sided [0.0045 to 0.0295] — Difference = Path Length per second (Typical) - Path Length per second (Atypical)

8. Primary Outcome: Center of Pressure, Path Length Per Second - Lion Toy (Motor Control Outcome)
Description: Body movement (center of pressure) on a mat, in terms of path length per minute. Early postural control (measured by center of pressure) was investigated to distinguish infants with future impairment in motor control from their typically developing peers. Lower path length is representative of greater postural control. The data analyzed was the condition where infant supine movement on the mat for up to two minutes with lion toy. Path length was measured in distance with time normalized to 1 minute.
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per second (cm/sec)
Arm/Group | Infants - Typical Development | Infants - Atypical Development
Number analyzed (Participants) | 11 | 4
centimeters per second (cm/sec) | 0.0335 (0.0113) | 0.0416 (0.0025)
Statistical Analysis 1: Comparison: Infants - Typical Development vs Infants - Atypical Development; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.6782, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = 0.0066, 95% CI 2-sided [-0.0059 to 0.0191] — Difference = Path Length per second (Typical) - Path Length per second (Atypical)

9. Primary Outcome: Center of Pressure, Standard Deviation (Y) - No Toy (Birth Status)
Description: Body movement (center of pressure) on a mat, in terms of standard deviation Y. Early postural control (measured by center of pressure) was investigated to distinguish infants with future impairment in motor control from their typically developing peers. Lower path length is representative of greater postural control. The data analyzed was the condition where infant supine movement on the mat for up to two minutes without a toy. Path length was measured in distance with time normalized to 1 minute.
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per minute (cm/min)
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 8 | 7
centimeters per minute (cm/min)
  *StdDevY (Full-Term): number analyzed (Participants) | 8 | 0
  *StdDevY (Full-Term) | 1.863 (0.920) |
  *StdDevY (Pre-Term): number analyzed (Participants) | 0 | 7
  *StdDevY (Pre-Term) |  | 0.799 (0.502)
Statistical Analysis 1: Comparison: Full-Term Infants vs Pre-Term Infants; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.0479, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = 1.064, 95% CI 2-sided [0.006 to 2.122] — Difference = StdDevY (Full-Term) - StdDevY (Pre-Term)

10. Primary Outcome: Center of Pressure, Standard Deviation (Y) - Elephant Toy (Birth Status)
Description: Body movement (center of pressure) on a mat, in terms of standard deviation Y. Early postural control (measured by center of pressure) was investigated to distinguish infants with future impairment in motor control from their typically developing peers. Lower path length is representative of greater postural control. The data analyzed was the condition where infant supine movement on the mat for up to two minutes with elephant toy. Path length was measured in distance with time normalized to 1 minute.
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per minute (cm/min)
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 8 | 7
centimeters per minute (cm/min) | 1.520 (0.710) | 1.159 (1.001)
Statistical Analysis 1: Comparison: Full-Term Infants vs Pre-Term Infants; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.9947, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = 0.278, 95% CI 2-sided [-0.921 to 1.477] — Difference = StdDevY (Full-Term) - StdDevY (Pre-Term)

11. Primary Outcome: Center of Pressure, Standard Deviation (Y) - Orangutan Toy (Birth Status)
Description: Body movement (center of pressure) on a mat, in terms of standard deviation Y. Early postural control (measured by center of pressure) was investigated to distinguish infants with future impairment in motor control from their typically developing peers. Lower path length is representative of greater postural control. The data analyzed was the condition where infant supine movement on the mat for up to two minutes with orangutan toy. Path length was measured in distance with time normalized to 1 minute.
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per minute (cm/min)
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 8 | 7
centimeters per minute (cm/min) | 1.857 (0.981) | 0.890 (0.540)
Statistical Analysis 1: Comparison: Full-Term Infants vs Pre-Term Infants; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.2614, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = 0.835, 95% CI 2-sided [-0.274 to 1.945] — Difference = StdDevY (Full-Term) - StdDevY (Pre-Term)

12. Primary Outcome: Center of Pressure, Standard Deviation (Y) - Lion Toy (Birth Status)
Description: Body movement (center of pressure) on a mat, in terms of standard deviation Y. Early postural control (measured by center of pressure) was investigated to distinguish infants with future impairment in motor control from their typically developing peers. Lower path length is representative of greater postural control. The data analyzed was the condition where infant supine movement on the mat for up to two minutes with lion toy. Path length was measured in distance with time normalized to 1 minute.
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per minute (cm/min)
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 8 | 7
centimeters per minute (cm/min) | 2.046 (0.658) | 0.738 (0.285)
Statistical Analysis 1: Comparison: Full-Term Infants vs Pre-Term Infants; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.0314, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = 1.176, 95% CI 2-sided [0.066 to 2.286] — Difference = StdDevY (Full-Term) - StdDevY (Pre-Term)

13. Primary Outcome: Center of Pressure, Standard Deviation (Y) - No Toy (Motor Control Outcome)
Description: as for outcome 9
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per second (cm/sec)
Arm/Group | Infants - Typical Development | Infants - Atypical Development
Number analyzed (Participants) | 11 | 4
centimeters per second (cm/sec) | 1.6920 (0.9442) | 0.6177 (0.3032)
Statistical Analysis 1: Comparison: Infants - Typical Development vs Infants - Atypical Development; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.0958, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = -1.074, 95% CI 2-sided [-2.255 to 0.1059] — Difference = StdDevY (Typical) - StdDevY (Atypical)

14. Primary Outcome: Center of Pressure, Standard Deviation (Y) - Elephant Toy (Motor Control Outcome)
Description: as for outcome 10
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per second (cm/sec)
Arm/Group | Infants - Typical Development | Infants - Atypical Development
Number analyzed (Participants) | 11 | 4
centimeters per second (cm/sec) | 1.3491 (0.7232) | 1.6428 (1.7433)
Statistical Analysis 1: Comparison: Infants - Typical Development vs Infants - Atypical Development; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.9660, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = 0.5248, 95% CI 2-sided [-1.1243 to 2.1739] — Difference = StdDevY (Typical) - StdDevY (Atypical)

15. Primary Outcome: Center of Pressure, Standard Deviation (Y) - Orangutan Toy (Motor Control Outcome)
Description: as for outcome 11
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per second (cm/sec)
Arm/Group | Infants - Typical Development | Infants - Atypical Development
Number analyzed (Participants) | 11 | 4
centimeters per second (cm/sec) | 1.5857 (1.0106) | 1.0820 (0.6662)
Statistical Analysis 1: Comparison: Infants - Typical Development vs Infants - Atypical Development; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.9462, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = -0.4198, 95% CI 2-sided [-1.6278 to 0.7882] — Difference = StdDevY (Typical) - StdDevY (Atypical)

16. Primary Outcome: Center of Pressure, Standard Deviation (Y) - Lion Toy (Motor Control Outcome)
Description: as for outcome 12
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters per second (cm/sec)
Arm/Group | Infants - Typical Development | Infants - Atypical Development
Number analyzed (Participants) | 11 | 4
centimeters per second (cm/sec) | 1.8048 (0.7578) | 0.6503 (0.2535)
Statistical Analysis 1: Comparison: Infants - Typical Development vs Infants - Atypical Development; Test type: Superiority — Two-Factor ANOVA in repeated measures; p = 0.1129, ANOVA — The threshold for statistical significance was p = 0.05; p Values were adjusted for multiple comparisons using Tukey-Kramer tests; Mean Difference (Net) = -1.0705, 95% CI 2-sided [-2.2785 to 0.1375] — Difference = StdDevY (Typical) - StdDevY (Atypical)

17. Primary Outcome: Toy Interaction (Elephant Toy) - Grasp/Touch/Kick/Mouth Time
Description: Time duration (in seconds) of infant interaction with the Elephant toy. Time spent in voluntary motor (feet and hand) interactions with the toy, analyzing grasp/touch/kick/mouth time. The data analyzed was the condition where the elephant toy was suspended within arm reach above the supine infant for approximately 120 seconds. The median and IQR measure the number of seconds the infant spent interacting with the toy. For numbers that were reported (0,0), those infants had no reaction and spent no time interacting with the toy. Toy interaction time ranged from 0-120 seconds.
Time Frame: 1 session, approximately 120 seconds during session 1 for the Elephant toy
Population: 13 excluded from enrolled 36: 2 infants were excluded from Toy Interaction analysis due to procedural adjustments.
  5 were excluded from Toy Interaction analysis due to procedural inconsistencies.
  6 were excluded from Toy Interaction analysis from unusable data (infants were either crying or crawling/rolling off the gym).
Measure: Median (Inter-Quartile Range); unit: second (s)
Groups:
- Full-Term Infants; Pre-Term Infants: Two populations will be involved in testing in the SmarToyGym: 1. Full-term infants (born at a gestational age of > 37 weeks) between 3 months and 11 months of age. 2. Pre-term infants (born at a gestational age < 36 weeks) between 3 months and 11 months of age.
  SmarToyGym: We aim to develop a SmarToyGym where sensitized, wireless toys are strategically hung and placed within reach of infants to elicit toy-oriented body and arm/hand movements. Each toy will be equipped with sensors capable of measuring the infant's grasping actions such as squeezing, pinching, tilting, etc.
  A low-cost 3D motion capture system will be used to collect video data and the infants' reaching and body kinematics in response to the toys. A pressure mat will be used to measure postural changes to detect weight shifts, rolling, crawling and other movements away from the initial posture.
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 14 | 9
second (s) | 90.7 [0 to 190.7] | 0 [0 to 0]

18. Primary Outcome: Toy Interaction (Orangutan Toy) - Grasp/Touch/Kick/Mouth Time
Description: Time duration (in seconds) of infant interaction with the Orangutan toy. Time spent in voluntary motor (feet and hand) interactions with the toy, analyzing grasp/touch/kick/mouth time. The data analyzed was the condition where the orangutan toy was suspended within arm reach above the supine infant for approximately 120 seconds. The median and IQR measure the number of seconds the infant spent interacting with the toy. For numbers that were reported (0,0), those infants had no reaction and spent no time interacting with the toy. Toy interaction time ranged from 0-120 seconds.
Time Frame: 1 session, approximately 120 seconds during session 1 for the Orangutan toy
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: seconds (s)
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 14 | 9
seconds (s) | 69.3 [26.3 to 240.1] | 27.9 [0 to 30.4]

19. Primary Outcome: Toy Interaction (Lion Toy) - Grasp/Touch/Kick/Mouth Time
Description: Time duration (in seconds) of infant interaction with the Lion toy. Time spent in voluntary motor (feet and hand) interactions with the toy, analyzing grasp/touch/kick/mouth time. The data analyzed was the condition where the lion toy was suspended within foot reach above the supine infant for approximately 120 seconds. The median and IQR measure the number of seconds the infant spent interacting with the toy. For numbers that were reported (0,0), those infants had no reaction and spent no time interacting with the toy. Toy interaction time ranged from 0-120 seconds.
Time Frame: 1 session, approximately 120 seconds during session 1 for the Lion toy
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: seconds (s)
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 14 | 9
seconds (s) | 2.2 [0 to 25.7] | 0 [0 to 0]

20. Primary Outcome: Toy Interaction (Elephant Toy) - Gaze Time
Description: Time duration (in seconds) of infant interaction with the Elephant toy. Time spent gazing at the toy. The data analyzed was the condition where the elephant toy was suspended within arm reach above the supine infant for approximately 120 seconds. The median and IQR measure the number of seconds the infant spent gazing at the toy. For numbers that were reported (0,0), those infants had no reaction and spent no time gazing at the toy. Toy interaction time ranged from 0-120 seconds.
Time Frame: 1 session, approximately 120 seconds during session 1 for the Elephant toy
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: seconds (s)
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 14 | 9
seconds (s) | 59.6 [22.6 to 71.4] | 0 [0 to 4.7]

21. Primary Outcome: Toy Interaction (Orangutan Toy) - Gaze Time
Description: Time duration (in seconds) of infant interaction with the Orangutan toy. Time spent gazing at the toy. The data analyzed was the condition where the orangutan toy was suspended within arm reach above the supine infant for approximately 120 seconds. The median and IQR measure the number of seconds the infant spent gazing at the toy. For numbers that were reported (0,0), those infants had no reaction and spent no time gazing at the toy. Toy interaction time ranged from 0-120 seconds.
Time Frame: 1 session, approximately 120 seconds during session 1 for the Orangutan toy
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: seconds (s)
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 14 | 9
seconds (s) | 83.5 [60.3 to 96.9] | 44.8 [37.6 to 84]

22. Primary Outcome: Toy Interaction (Lion Toy) - Gaze Time
Description: Time duration (in seconds) of infant interaction with the Lion toy. Time spent gazing at the toy. The data analyzed was the condition where the lion toy was suspended within foot reach above the supine infant for approximately 120 seconds. The median and IQR measure the number of seconds the infant spent gazing at the toy. For numbers that were reported (0,0), those infants had no reaction and spent no time gazing at the toy. Toy interaction time ranged from 0-120 seconds.
Time Frame: 1 session, approximately 120 seconds during session 1 for the Lion toy
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: seconds (s)
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 14 | 9
seconds (s) | 21.7 [7.3 to 57.5] | 0 [0 to 0]

23. Primary Outcome: Number of Occurrences of Elephant Toy Interactions
Description: Frequency of infant interactions with the Elephant toy. Frequency of mouthing, grasping, hand touch, foot touch, and kicking with the toy. The data analyzed was the condition where the elephant toy was suspended within arm reach above the supine infant for approximately 120 seconds. The median and IQR measure the number of occurrences the infant had interacting with the toy. For numbers that were reported (0,0), those infants had no reaction and spent no time interacting with the toy.
Time Frame: 1 session, approximately 120 seconds during session 1 for the Elephant toy
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: occurrences
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 14 | 9
occurrences | 22.5 [0 to 32] | 0 [0 to 2]

24. Primary Outcome: Number of Occurrences of Orangutan Toy Interactions
Description: Frequency of infant interactions with the Orangutan toy. Frequency of mouthing, grasping, hand touch, foot touch, and kicking with the toy. The data analyzed was the condition where the orangutan toy was suspended within arm reach above the supine infant for approximately 120 seconds. The median and IQR measure the number of occurrences the infant had interacting with the toy. For numbers that were reported (0,0), those infants had no reaction and spent no time interacting with the toy.
Time Frame: 1 session, approximately 120 seconds during session 1 for the Orangutan toy
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: occurrences
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 14 | 9
occurrences | 7 [5 to 16] | 7 [0 to 13]

25. Primary Outcome: Number of Occurrences of Lion Toy Interactions
Description: Frequency of infant interactions with the Lion toy. Frequency of mouthing, grasping, hand touch, foot touch, and kicking with the toy. The data analyzed was the condition where the lion toy was suspended within foot reach above the supine infant for approximately 120 seconds. The median and IQR measure the number of occurrences the infant had interacting with the toy. For numbers that were reported (0,0), those infants had no reaction and spent no time interacting with the toy.
Time Frame: 1 session, approximately 120 seconds during session 1 for the Lion toy
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: occurrences
Arm/Group | Full-Term Infants | Pre-Term Infants
Number analyzed (Participants) | 14 | 9
occurrences | 1 [0 to 19] | 0 [0 to 0]

26. Secondary Outcome: Wrist Position
Description: Kinematic planar (x, y) representation of wrist position (in l) based on pose captured from a single camera and through machine learning. Right and left arm wrist position were measured. Wrist position is reported in pixels from the camera data and normalization of data (units of measure is represented as pixels per length of trunk, normalized units with respect to trunk length). A positive value indicates the movement of arm upwards, and a negative value indicates the movement of arm downwards, with respect to the baseline.
  The camera data analyzed was the condition where infant supine movement on the mat for up to two minutes (without a toy). The camera was in a fixed position above the infant.
Time Frame: 1 session, about 1 hour in length
Population: 13 full-term, 6 pre-term. 17 excluded from enrolled 36: 5 were excluded from wrist/ankle analysis due to procedural adjustments. 7 were excluded from wrist/ankle analysis due to missing BINS score data. 2 were excluded from wrist/ankle analysis due to unusable data (infants were sitting during the video, which prevented successful pose estimation).
  3 were excluded from wrist/ankle analysis due to missing video data.
Measure: Median (Standard Deviation); unit: pixels per normalized trunk length
Groups:
- Low-Risk Infants; Moderate-Risk Infants; High-Risk Infants: Two populations will be involved in testing in the SmarToyGym: 1. Full-term infants (born at a gestational age of > 37 weeks) between 3 months and 11 months of age. 2. Pre-term infants (born at a gestational age < 36 weeks) between 3 months and 11 months of age.
  The risk of neuromotor dysfunction was classified by the BINS test (low, moderate, high) computed at corrected aged for preterm infants and chronological age for full-term infants.
  SmarToyGym: We aim to develop a SmarToyGym where sensitized, wireless toys are strategically hung and placed within reach of infants to elicit toy-oriented body and arm/hand movements. Each toy will be equipped with sensors capable of measuring the infant's grasping actions such as squeezing, pinching, tilting, etc.
  A low-cost 3D motion capture system will be used to collect video data and the infants' reaching and body kinematics in response to the toys. A pressure mat will be used to measure postural changes to detect weight shifts, rolling, crawling and other movements away from the initial posture.
Arm/Group | Low-Risk Infants | Moderate-Risk Infants | High-Risk Infants
Number analyzed (Participants) | 5 | 9 | 5
pixels per normalized trunk length
  Wrist Position, x | 0.008 (0.031) | 0.088 (0.239) | -0.044 (0.146)
  Wrist Position, y | 0.370 (0.229) | 0.268 (0.217) | 0.224 (0.185)

27. Secondary Outcome: Ankle Position
Description: Kinematic planar (x, y) representation of ankle position (in l) based on pose captured from a single camera and through machine learning. Right and left arm ankle position were measured. Ankle position is reported in pixels from the camera data and normalization of data (units of measure is represented as pixels per length of trunk, normalized units with respect to trunk length). A positive value indicates the movement of leg upwards, and a negative value indicates the movement of leg downwards, with respect to the baseline.
  The camera data analyzed was the condition where infant supine movement on the mat for up to two minutes (without a toy). The camera was in a fixed position above the infant.
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 26
Measure: Median (Standard Deviation); unit: pixels per normalized trunk length
Arm/Group | Low-Risk Infants | Moderate-Risk Infants | High-Risk Infants
Number analyzed (Participants) | 5 | 9 | 5
pixels per normalized trunk length
  Ankle Position, x | -0.018 (0.190) | 0.017 (0.176) | -0.056 (0.097)
  Ankle Position, y | 1.580 (0.076) | 1.472 (0.094) | 1.348 (0.389)

28. Secondary Outcome: Wrist Velocity
Description: Kinematic (x, y) representation of wrist movement (in l/s) based on pose captured from a single camera and through machine learning. Right and left arm wrist movement were measured. Wrist movement is reported in pixels from the camera data and normalization of data (units of measure is represented as pixels per length of trunk, normalized units with respect to trunk length). A positive value indicates the movement of arm upwards, and a negative value indicates the movement of arm downwards, with respect to the baseline.
  The camera data analyzed was the condition where infant supine movement on the mat for up to two minutes (without a toy). The camera was in a fixed position above the infant.
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 26
Measure: Median (Standard Deviation); unit: pixels (per trunk length) per second
Arm/Group | Low-Risk Infants | Moderate-Risk Infants | High-Risk Infants
Number analyzed (Participants) | 5 | 9 | 5
pixels (per trunk length) per second
  Wrist Velocity, x | 0.034 (0.014) | 0.048 (0.017) | 0.048 (0.023)
  Wrist Velocity, y | 0.035 (0.016) | 0.045 (0.019) | 0.054 (0.023)

29. Secondary Outcome: Ankle Velocity
Description: Kinematic (x, y) representation of ankle movement (in l/s) based on pose captured from a single camera and through machine learning. Right and left ankle movement were measured. Ankle movement is reported in pixels from the camera data and normalization of data (units of measure is represented as pixels per length of trunk, normalized units with respect to trunk length). A positive value indicates the movement of leg upwards, and a negative value indicates the movement of leg downwards, with respect to the baseline.
  The camera data analyzed was the condition where infant supine movement on the mat for up to two minutes (without a toy). The camera was in a fixed position above the infant.
Time Frame: 1 session, about 1 hour in length
Population: as for outcome 26
Measure: Median (Standard Deviation); unit: pixels (per trunk length) per second
Arm/Group | Low-Risk Infants | Moderate-Risk Infants | High-Risk Infants
Number analyzed (Participants) | 5 | 9 | 5
pixels (per trunk length) per second
  Ankle Velocity, x | 0.052 (0.020) | 0.072 (0.029) | 0.067 (0.042)
  Ankle Velocity, y | 0.041 (0.018) | 0.067 (0.039) | 0.062 (0.046)

ADVERSE EVENTS:
Time Frame: 1 hour participation sessions, over 8 months
Arm/Group | Full-Term Infants | Pre-Term Infants
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/10
Other Adverse Events (participants affected / at risk) | 0/26 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT02813889/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT02813889/ICF_001.pdf